CLINICAL TRIAL: NCT06448780
Title: Dose Optimization of Caffeine in Neonates With Hypoxic-Ischemic Encephalopathy
Brief Title: Dose Optimization of Caffeine for HIE
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 24-0654; 1K23HD111623-01 (NIH)
Record Dates: First submitted 2024-06-03; First posted 2024-06-07 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Hypoxic-Ischemic Encephalopathy
Keywords: caffeine citrate
MeSH Terms: conditions — Hypoxia-Ischemia, Brain | interventions — caffeine citrate

STUDY DESIGN:
Intervention Model Description: The first cohort of 8 infants will receive a lower loading dose of caffeine. Following a safety review, an additional 8 infants will receive a higher loading dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Lower loading dose (20 mg/kg) (Active Comparator): Within 24 hours after delivery, participants will receive a loading dose of 20 mg/kg caffeine citrate IV.
  Interventions: Drug: Caffeine citrate 20 mg/kg
- Higher loading dose (30 mg/kg) (Active Comparator): Within 24 hours after delivery, participants will receive a loading dose of 30 mg/kg caffeine citrate IV.
  Interventions: Drug: Caffeine citrate 30 mg/kg

INTERVENTIONS:
Drug: Caffeine citrate 20 mg/kg — Following loading dose of 20 mg/kg of caffeine citrate IV, participants will receive 2 daily doses of 10 mg/kg caffeine citrate IV.
  Other Names: Cafcit
  Arms: Lower loading dose (20 mg/kg)
Drug: Caffeine citrate 30 mg/kg — Following loading dose of 30 mg/kg of caffeine citrate IV, participants will receive 2 daily doses of 10 mg/kg caffeine citrate IV.
  Other Names: Cafcit
  Arms: Higher loading dose (30 mg/kg)

SUMMARY:
This is a phase Ib, open-label, dose-validating and safety study of caffeine in neonates with hypoxic-ischemic encephalopathy (HIE) undergoing therapeutic hypothermia.

DETAILED DESCRIPTION:
In a previous phase I trial (NCT03913221), the investigators characterized the pharmacokinetics (PK) of caffeine in the setting of HIE and therapeutic hypothermia using a population PK model. This is an open-label study of caffeine citrate in neonates with HIE to validate the population PK model and determine optimal dosing for HIE.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent from parent or guardian
* ≥ 36 weeks gestational age at birth
* Receiving therapeutic hypothermia for a diagnosis of HIE
* Intravenous (IV) access
* Postnatal age < 24 hours

Exclusion Criteria:

* Receiving > 1 anti-epileptic drug for seizures
* Sustained (>4 hours) heart rate > 180 beats per minute
* Known major congenital anomaly

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 16 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Apparent Caffeine Clearance | 7 samples will be collected after the first dose of study drug and up to 72 hours after final dose of study drug
  Clearance is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Caffeine concentrations will be used to calculate population estimates of caffeine clearance, with inter-individual variabilty and residual variabilty .
Volume of Distribution of Caffeine | 7 samples will be collected after the first dose of study drug and up to 72 hours after final dose of study drug
  Caffeine concentrations will be used to calculate population estimates of volume of distribution with inter-individual variability and residual variability.

SECONDARY OUTCOMES:
Number of Participants with Pre-Specified Adverse Events | From the first dose of caffeine to 7 days following the final dose.
  Safety will be determined by the number of participants with the following: seizures requiring > 1 anti-epileptic drug, necrotizing enterocolitis defined as Bell Stage II or higher, hypoglycemia defined as point-of-care blood glucose < 30 mg/dL, and hyperglycemia defined as point-of-care blood glucose >200 mg/dL.
Number of Participants with Abnormal MRI Brain Finding Score | During initial hospitalization, typically 3-5 postnatal days
  Preliminary effectiveness assessed using the NICHD Neonatal Research Network MRI scoring system that categorizes severity of brain injury in the Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. Abnormal MRI is defined as any score >0.
  * Score 0: Normal MRI
  * Score 1A: Minimal cerebral lesions only with involvement of basal ganglia, thalamus
  * Score 1B: Extensive cerebral lesions
  * Score 2A: Basal ganglia thalamic, anterior or posterior limb of internal capsule, or watershed infarction
  * Score 2B: 2A with cerebral lesions
  * Score 3: Hemispheric devastation
Number of Participants with Death or Neurodevelopmental Impairment | 18-24 months of age
  Preliminary effectiveness assessed based on death or neurodevelopmental impairment defined as: diagnosis of cerebral palsy, hearing impairment requiring hearing aids, blindness, or cognitive, language, or motor score < 85 on the Bayley Scales of Infant and Toddler Development- Fourth Edition.

CONTACTS AND LOCATIONS:
Overall Officials: Wesley M Jackson, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- The University of North Carolina at Chapel Hill Newborn Critical Care Center, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual data that supports the results will be shared beginning 9 to 36 months following publication provided the investigator who proposes to use the data has approval from an Institutional Review Board (IRB), Independent Ethics Committee (IEC), or Research Ethics Board (REB), as applicable, and executes a data use/sharing agreement with UNC.
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication.
Access Criteria: Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata.

REFERENCES:
- [Background] Shankaran S, McDonald SA, Laptook AR, Hintz SR, Barnes PD, Das A, Pappas A, Higgins RD; Eunice Kennedy Shriver National Institute of Child Health and Human Development Neonatal Research Network. Neonatal Magnetic Resonance Imaging Pattern of Brain Injury as a Biomarker of Childhood Outcomes following a Trial of Hypothermia for Neonatal Hypoxic-Ischemic Encephalopathy. J Pediatr. 2015 Nov;167(5):987-93.e3. doi: 10.1016/j.jpeds.2015.08.013. Epub 2015 Sep 16. PMID 26387012
- [Background] Selewski DT, Charlton JR, Jetton JG, Guillet R, Mhanna MJ, Askenazi DJ, Kent AL. Neonatal Acute Kidney Injury. Pediatrics. 2015 Aug;136(2):e463-73. doi: 10.1542/peds.2014-3819. Epub 2015 Jul 13. PMID 26169430
- [Background] Jackson W, Gonzalez D, Greenberg RG, Lee YZ, Laughon MM. A phase I trial of caffeine to evaluate safety in infants with hypoxic-ischemic encephalopathy. J Perinatol. 2024 Apr;44(4):508-512. doi: 10.1038/s41372-023-01752-y. Epub 2023 Aug 16. PMID 37587184